CLINICAL TRIAL: NCT04366297
Title: Intraosseous Versus Intravenous Access During COVID-19 Patients Performed by Paramedics Wearing Level C Personal Protective Equipment. A Multi-center Prospective Randomized Crossover Single-blinded Simulation Trial
Brief Title: Intravascular Access of COVID-19 Patient Under Personal Protective Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Collaborators: Poznan University of Medical Sciences (Other); Medical University of Bialystok (Other); Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Assoc Prof PhD, Lazarski University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IO_PPE_MS_1
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Arrest; Emergencies
Keywords: intravascular access; COVID-19; personal protective equipment; medical simulation
MeSH Terms: conditions — Heart Arrest; Emergencies; COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Intravenous Cannula) (Experimental): obtaining intravascular access using a ready standard intravenous cannula
  Interventions: Device: Intravenous access
- IO access using NIO® set (Experimental): receive an IO line in the proximal tibia localization. IO lines are placed using an FDA-approved device called an NIO®.
  Interventions: Device: Intraosseous access

INTERVENTIONS:
Device: Intravenous access — obtaining intravascular access using a standard intravenous cannula
  Other Names: IV
  Arms: Standard of Care (Intravenous Cannula)
Device: Intraosseous access — obtaining intravascular access using a ready intravenous NIO needle set
  Other Names: IO
  Arms: IO access using NIO® set

SUMMARY:
The current COVID-19 pandemic, this is especially since the transmission of SARS-CoV-2 is thought to occur mainly through respiratory droplets generated by coughing and sneezing, by direct contact with contaminated surfaces and because in a large number of patients COVID-19 disease may be asymptomatic. As recommended by the CDC medical personnel should be equipped with full personal protective equipment (PPE) for AGP in contact with suspected/confirmed COVID-19 patient. Therefore, it is reasonable to search for the most effective methods of intravascular access in those conditions.

ELIGIBILITY:
Inclusion Criteria:

* paramedic
* consent voluntary participation in the study
* none experience in resuscitation with personal protective equipment

Exclusion Criteria:

* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
successful rate of first intravascular access attempt | 1 day
  successful placement of intravascular device

SECONDARY OUTCOMES:
time to successful access | 1 day
number of attempts to successful access | 1 day
  number of attempts to successful access
time to infusion | 1 day
  time to therapy including but not limited to time to fluids, antibiotics, and antiarrythmics
complication rates | 1 day
  complication rates
ease of use | 1 day
  self-reported percentage the vocal cord visualization. A 100% score is a extremely difficult procedure. A Ease of use score of 1% means that procedure is extremely easy
Preferred intravascular access method | 1 day
  participants were asked which method of intravascular access they would prefer in a real-life resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Smereka, PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Lazarski Univeristy, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
the investigators will add data into manuscript

REFERENCES:
- [Background] Smereka J, Szarpak L, Filipiak KJ, Jaguszewski M, Ladny JR. Which intravascular access should we use in patients with suspected/confirmed COVID-19? Resuscitation. 2020 Jun;151:8-9. doi: 10.1016/j.resuscitation.2020.04.014. Epub 2020 Apr 15. No abstract available. PMID 32304800